CLINICAL TRIAL: NCT04211545
Title: A Phase 1, Open-label Study to Assess the Single Dose Pharmacokinetics and Relative Bioavailability of a Test Capsule Formulation of CC-92480 Compared to a Reference CC 92480 Capsule Formulation and the Effect of a Proton Pump Inhibitor on the Pharmacokinetics of CC 92480 From Test and Reference Formulations in Healthy Subjects
Brief Title: Relative Bioavailability and PPI Effects of CC-92480 Test and Reference Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CC-92480-CP-002; U1111-1242-7394 (Other: WHO)
Record Dates: First submitted 2019-12-24; First posted 2019-12-26 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Healthy Volunteer
Keywords: Healthy Subjects; CC-92480; Pharmacokinetics
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of CC-92480 and Rabeprazole (Experimental): Test Formulation CC-92480 and Reference Formulation will be administered orally at 1.6 mg. Rabeprazole will be administered orally at 40 mg.
  Interventions: Drug: Rabeprazole; Drug: CC-92480

INTERVENTIONS:
Drug: Rabeprazole — Rabeprazole
Drug: CC-92480 — CC-92480

SUMMARY:
This is a Phase 1, open-label, randomized, four-period, crossover study in healthy females of nonchildbearing potential and male subjects - to be conducted at a single center in the United States.

The study will consist of a screening phase, a baseline phase, four treatment periods, and a follow-up phone call. The 4 treatment periods are divided into two pairs (Period 1 and 2 and Period 3 and 4), potentially separated by an intermission during which subjects will be discharged from the research unit: Periods 1 and 2 support relative bioavailability (RBA) estimation, while Periods 3 and 4 support estimation of PPI effects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study (partial):

1. Must understand and voluntarily sign a written informed consent form (ICF) prior to any study-related assessments/procedures being performed.
2. Must be able to communicate with the Investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
3. Healthy adult male or female of any race, between 18 to 55 years of age (inclusive) at the time of signing the ICF, and in good health as determined by the screening history and PE.
4. For males:

   1. Practice true abstinence (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 3 months following investigational product discontinuation, even if he has undergone a successful vasectomy.
   2. Agree to use barrier contraception not made of natural (animal) membrane (eg, latex or polyurethane condoms are acceptable) when engaging in sexual activity with a female of childbearing potential (FCBP) 1 while on study medication, and for at 3 months after the last dose of study medication.
5. Must have a body mass index between 18 and 33 kg/m2 (inclusive) at the time of signing the ICF.
6. Clinical laboratory test results must be within the respective reference ranges; or if not, the results be clinically insignificant according to the Investigator's medical judgement.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. History of any clinically significant and relevant neurological, GI, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders as determined by the Investigator.
2. Exposure to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
3. Use of tobacco - or nicotine-containing products within 3 months prior to Day -1 (Period 1 for Part 2).
4. Vaccination within 30 days of first dose administration or plans to receive vaccination within 30 days after dosing.
5. Subjects with active hepatitis and HIV
6. Use of any nonprescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration.
7. Use of CYP3A inducers and inhibitors (including St. John's Wort) within 30 days of the first dose administration.
8. Any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion (ADME), eg, bariatric procedure. Appendectomy and cholecystectomy are acceptable. Prior procedures of unclear ADME significance should be reviewed with the Sponsor's Medical Monitor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - AUC0-∞ (Reference Formulation) | Up to 5 days
  Area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics - AUC0-∞ (Test Formulation) | Up to 5 days
  Area under the plasma concentration-time curve from time zero to the last observable concentration at time t

SECONDARY OUTCOMES:
Pharmacokinetics -Cmax (Reference Formulation) | Day 1
  Maximum plasma concentration
Pharmacokinetics - Cmax (Test Formulation) | Day 1
  Maximum plasma concentration
Pharmacokinetics - AUC0-t (Reference Formulation) | Up to 5 days
  Area under the plasma concentration-time curve from time zero to the last observable concentration at time t
Pharmacokinetics - AUC0-t (Test Formulation) | Up to 5 days
  Area under the plasma concentration-time curve from time zero to the last observable concentration at time t
Pharmacokinetics -Tmax (Reference Formulation) | Day 1
  Time to peak (maximum) plasma concentration
Pharmacokinetics -Tmax (Test Formulation) | Day 1
  Time to peak (maximum)plasma concentration
Pharmacokinetics - CL/F (Reference Formulation) | Up to 5 days
  Apparent total plasma clearance
Pharmacokinetics - CL/F (Test Formulation) | Up to 5 days
  Apparent total plasma clearance
Pharmacokinetics - Vz/F (Reference Formulation) | Up to 5 days
  Apparent volume of distribution
Pharmacokinetics - Vz/F (Test Formulation) | Up to 5 days
  Apparent volume of distribution
Pharmacokinetics - t1/2 (Reference Formulation) | Up to 5 days
  Terminal elimination half-life
Pharmacokinetics - t1/2 (Test Formulation) | Up to 5 days
  Terminal elimination half-life
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values (as specified by the criteria in Section 10.3), regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Carayannopoulos, MD, Study Director — Celgene
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Wu F, Liu L, Gaudy A, Wang X, Carayannopoulos L, Pourdehnad M, Lamba M. Model based assessment of food and acid reducing agent effects on oral absorption of mezigdomide (CC-92480), a novel cereblon E3 ligase modulator. CPT Pharmacometrics Syst Pharmacol. 2023 Oct;12(10):1473-1484. doi: 10.1002/psp4.13024. Epub 2023 Sep 13. PMID 37705327